CLINICAL TRIAL: NCT06688383
Title: "Anastomotic Leakage After Right Hemicolectomy for Cancer, a Prospective Multicenter Study of SICO-CC Network." (AL RIGHT).
Brief Title: Anastomotic Leakage After Right Hemicolectomy for Cancer, a Prospective Multicenter Study of SICO-CC Network
Acronym: ALRIGHT
Status: Recruiting | Type: Observational
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Rossella Reddavid, MD, PHD, San Luigi Gonzaga Hospital
Other Study IDs: ALRIGHT01
Record Dates: First submitted 2024-10-17; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Anastomotic Leak Large Intestine; Right Colon Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a nationwide prospective observational study to assess the overall clinical anastomotic leakage rate after right hemicolectomy for cancer, to detect the independent risk factors for AL, and to develop a clinical prediction model to estimates of the probability of the occurrence of an AL after surgery. Since this is a multicenter prospective study, the Division of Surgical Oncology and Digestive Surgery from the University of Turin, Department of Oncology, AOU San Luigi Gonzaga di Orbassano will be the Coordinator Center of the study, Ethics committee approves will be requested before the implementation of this study.

Italian high-volume colorectal surgery centers members of SICO (The Italian Society of Oncological Surgery) have agreed to participate as collaborators of this study, notification and revision from their local ethics committee will be requested as well. A certified general surgeon with a large experience in the preoperative, operative, and postoperative management of patients with colorectal cancer has been identified to coordinate the study in each center. Id information of the potential collaborators is specified in the section "Trial Setting". Once the study is activated, eligible patients (or a representative) must provide written, informed consent before any study procedures occur. No intervention or modification of the habitual clinical practice is planned All data will enter into a database provided by the promoting center. There are three main sections of data collection for each patient:

* Preoperative: baseline, disease and demographics.
* Operative: details about the surgery, anastomosis construction and enterotomy closure.
* Follow-up: outcomes data about the early (within 30 postoperative day) and late postoperative course (31 th - 60th postoperative day) and pathology report. The definition of AL is based on the presence of clinical signs (pain, fever, tachycardia, peritonitis, feculent or enteric drainage, purulent drainage, postoperative ileus, abscess, septicemia, and/or organ failure) with radiographic signs (fluid collections, gas containing collections at CT scan) suggestive of AL and-or intraoperative or autopsy findings (gross enteric spillage, anastomotic disruption). The absence of AL will be assumed by a normal postoperative course and the absence of symptoms suggestive of AL with or without radiologic confirmation.

ELIGIBILITY:
Inclusion Criteria:

* Patients from all participating centers older than 18 years, males or females, with the diagnosis of primary right colon cancer including the cecum, ascendent, liver flexure, and proximal third of the transverse colon, in both emergency and elective settings, with the indication of RH, referred as to the resection of a portion of the distal ileum, cecum, ascending colon, and proximal to the mid-transverse colon, with intraperitoneal or extraperitoneal primary handsewn or mechanical ileocolic anastomosis by minimally invasive(robotic or laparoscopic) or open approach.

Exclusion Criteria:

* -Long steroid treatment for any cause.
* Right colon resection for benign disease.
* History of supra-mesocolic space radiotherapy.
* Inflammatory bowel disease (Crohn's disease and ulcerative colitis). No healthy volunteers are accepted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from all participating centers older than 18 years, males or females, with the diagnosis of primary right colon cancer including the cecum, ascendent, liver flexure, and proximal third of the transverse colon, in both emergency and elective settings, with the indication of RH, referred as to the resection of a portion of the distal ileum, cecum, ascending colon, and proximal to the mid-transverse colon, with intraperitoneal or extraperitoneal primary handsewn or mechanical ileocolic anastomosis by minimally invasive(robotic or laparoscopic) or open approach.
Sampling Method: Non-Probability Sample
Enrollment: 1839 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
overall rate of AL | from 1st to 30th postoperative day
  defined as the total cases of patients with clinical signs or symptoms of AL (pain, fever, tachycardia, peritonitis, feculent or enteric drainage, purulent drainage, postoperative ileus, abscess, septicemia, and/or organ failure), any radiological findings suggestive of AL (fluid collections, gas containing collections at CT scan) or intraoperative or autopsy findings (gross enteric spillage, anastomotic disruption), expressed in percentage. [time frame: from 1st to 30th postoperative day]. And identify the main associated factors through a multivariate model regression.

SECONDARY OUTCOMES:
overall morbidity | from 1st to 60 postoperative day
  The rate of overall morbidity in patients with and without AL. Refers to adverse events and complications following surgery and classified by Clavien Dindo score
operative mortality | within 30 postoperative days
  The rate of operative mortality in patients with and without AL. Operative mortality was defined as death that occurred within 30 days after the primary operation
Length of stay. | from date of surgery up to 200 days
  Total Length of stay. Defined as the length of an inpatient episode of care, calculated from the surgery day to the day of discharge and based on the number of nights spent in the hospital. Adding all the admissions episodes related and no related to AL
reoperation | from 1st to 60 postoperative day
  The rate of reoperation in patients with and without AL: defined of the total cases of patients submitted to secondary surgery for any direct untoward effect of the right colon resection

CONTACTS AND LOCATIONS:
Locations (1):
- San Luigi Gonzaga, Orbassano, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: Yes